CLINICAL TRIAL: NCT03118544
Title: REduction of Contrast Via DyeVert Used in CTO Procedures (REDUCe)
Brief Title: REduction of Contrast Via DyeVert Used in CTO Procedures
Acronym: REDUCe
Status: Terminated | Type: Observational
Why Stopped: Competing clinical trial priorities
Sponsor: Minneapolis Heart Institute Foundation (Other)
Collaborators: Osprey Medical, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: MinneapolisHIF
Record Dates: First submitted 2017-04-13; First posted 2017-04-18 (Actual); Last update posted 2018-05-17 (Actual); Status verified 2018-05

CONDITIONS: Chronic Total Occlusion of Coronary Artery
Keywords: Chronic Total Occlusion; Coronary Artery Disease; Percutaneous Coronary Intervention; CTO; PCI
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Patients undergoing CTO PCI: Evaluates the effect of the DyeVert System on contrast volume administration in patients undergoing clinically-indicated CTO PCI. The system allows monitoring and display of contrast volumes that are manually injected during the procedure which will be compared to physician entered contrast usage thresholds during angiographic procedures.
  Interventions: Device: DyeVert System

INTERVENTIONS:
Device: DyeVert System — The DyeVert System (Osprey Medical, Inc) consists of a Contrast Monitoring Wireless Display (CMW) and the DyeVert Plus Disposable Kit which is inclusive of a disposable single-use sterile Smart Syringe and DyeVert Plus Module.

SUMMARY:
The is an observational, prospective study to evaluate the effect of the DyeVert System on contrast volume administration in patients undergoing clinically-indicated chronic total occlusion (CTO) percutaneous coronary intervention (PCI)

DETAILED DESCRIPTION:
The DyeVert System is a disposable, FDA-approved device that interfaces with standard manifold systems to reduce the amount of contrast used in catheterization procedures, while maintaining fluoroscopic image opacity.

No study has assessed use of the system in CTO PCI. It would be expected that savings in CTO procedures may be less than non-CTO procedures due to catheter sizing and number of open guide injections required. Open guide injections through larger catheters do not provide for the as much resistance, therefore decreasing the need for contrast to be diverted

ELIGIBILITY:
Inclusion Criteria:

1. Subjects undergoing CTO PCI at each of the participating centers.
2. Contrast volume recorded during CTO PCI
3. Subjects included in the "Multicenter Registry of Chronic Total Occlusion Interventions" study (Allina IRB approval # 948134-1)

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients undergoing clinically-indicated chronic total occlusion (CTO) percutaneous coronary intervention (PCI)
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2017-03-26 (Actual); Primary Completion 2018-02-02 (Actual); Study Completion 2018-02-02 (Actual)

PRIMARY OUTCOMES:
Contrast volume administration during CTO PCI | During the CTO PCI procedure
  The hypothesis of the study is that use of the DyeVert System will result in lower contrast volume, determined through real-time monitoring with the DyeVert System.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Abbott Northwestern Hospital, Minneapolis, Minnesota
  - Minneapolis Heart Institute Foundation, Minneapolis, Minnesota
  - Minneapolis Heart Institute, Minneapolis, Minnesota

IPD SHARING:
Plan to Share IPD: No